CLINICAL TRIAL: NCT05097170
Title: Determining the Effect of Vital Parameters on Cerebral Oxygenation and Awareness During Ventricular Tachycardia Ablation
Brief Title: Cerebral Oxygenation and Awareness During VT Ablation
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Filiz Uzumcugil, Principal Investigator, Hacettepe University
Other Study IDs: GO-21/704
Record Dates: First submitted 2021-10-15; First posted 2021-10-28 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Cerebral Oxygenation
Keywords: cerebral oxygenation; ventricular tachycardia ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: patients under the age of 65
  Interventions: Procedure: NIRS during ventricular tachycardia ablation
- 2: patients above the age of 65
  Interventions: Procedure: NIRS during ventricular tachycardia ablation

INTERVENTIONS:
Procedure: NIRS during ventricular tachycardia ablation — NIRS: Near-infrared spectroscopy is a measurement technique that non-invasively and continuously monitors the balance between cerebral oxygen consumption and delivery.
  BIS: BIS is an electroencephalogram-derived parameter developed to monitor the hypnotic effects of anesthesia.
  Other Names: BIS during ventricular tachycardia ablation

SUMMARY:
It is aimed to examine the effect of the decrease in blood pressure that occurs during the ventricular tachycardia ablation process on cerebral oxygenation and awareness.

Patient's age, cardiac measurements (ejection fraction-EF), basal vital values, procedure time (especially activation and pacing mapping), and localization of the arrhythmia, may affect the NIRS and BIS response to blood pressure drop. In addition to the effects of patients' demographic information, cardiac capacity and procedure time on NIRS and BIS values (downtrend and duration), correlations of these values with other monitoring parameters (ETCO2 and SpO2) intended to be displayed.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18
* Patients who will undergo VT ablation
* Patients who want to participate in the study

Exclusion Criteria:

* Patients whose baseline values could not be obtained before induction
* Patients with severe neurological or psychiatric illness
* Patients who do not want to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients undergoing VT ablation procedure
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Near Infrared Spectrometer | perioperative (ventricular tachycardia ablation)
  cerebral oxygenation

SECONDARY OUTCOMES:
Bispectral Index | perioperative (ventricular tachycardia ablation)
  awareness

CONTACTS AND LOCATIONS:
Locations (1):
- Filiz Uzumcugil, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shivkumar K. Catheter Ablation of Ventricular Arrhythmias. N Engl J Med. 2019 Apr 18;380(16):1555-1564. doi: 10.1056/NEJMra1615244. No abstract available. PMID 30995375